CLINICAL TRIAL: NCT05581537
Title: Effect of Adding Systematic Desensitization to Goal Directed Paradigm on Risk of Falling in Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Heba Gaber, Assistant Lecturer, October 6 University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003940
Record Dates: First submitted 2022-07-17; First posted 2022-10-14 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (GA) (Experimental): receive systematic desensitization in addition to goal directed paradigm for eight weeks, Three sessions per week (1hour and half)
  Interventions: Other: Systematic Desensitization
- Control group (GB) (Experimental): receive goal directed paradigm for eight weeks, Three sessions per week (45 minutes)
  Interventions: Other: Systematic Desensitization

INTERVENTIONS:
Other: Systematic Desensitization — Systematic desensitization: 2 techniques
  1. Jacobson's technique (progressive muscle relaxation):
     It involves tensing and releasing muscles that progress through the body throughout focusing on mental relaxation throughout releasing muscle tension
  2. Guided imagery (vividly imagining):
  It includes 2 types of imagery training/mental practice (MP) which includes visual imagery is based on the sensory (visual) perception of the imagined movement and Kinesthetic imagery is based on sensory-motor information (proprioceptive). MP will be conducted in a quiet room, where each patient will be given detailed instructions to perform both visual and kinesthetic practice
  Other Names: Goal directed paradigm

SUMMARY:
Stroke is the leading cause of disability in the elderly . The most common manifestations of stroke are deficits in motor control that involve abnormal synergistic organization of movements, muscle weakness, sensory deficits, and loss of range of motion. Poor posture, which is one of its main symptoms, affects falls or injured falls.

Fear of falling is a psychological condition associated with balance disorders and fall risks after a stroke.

DETAILED DESCRIPTION:
Fear of falling can result in avoidance behavior, leading to inactivity and social isolation, and further exacerbate disability in stroke populations Systematic desensitization , one of cognitive behavior therapy (CBT), is a psychotherapeutic intervention designed to modify unrealistic beliefs that can contribute to negative emotions and behavior. Fear of falling could result from accurate perceptions of impaired balance ability and unrealistic beliefs about one's risk of falling.

Systematic desensitization may alter these self-defeating beliefs and thus reduce fear-avoidance behavior and the associated adverse consequences, such as limited social participation and is effective in reducing the fear of falling among older individuals Goal-directed training is an activity-based approach to therapy. Meaningful, client-selected goals are used to provide opportunities for problem solving and to indirectly drive the movements required to successfully meet the task demands. This is in contrast to interventions that focus on changing body functions. The approach is based on the dynamic systems motor control theory and occupation-based therapy models, which suggest that movement patterns emerge from the interaction between the person's abilities, environment and the goal. Four components provide the basis for goal-directed training: (1) selection of a meaningful goal; (2) analysis of baseline performance; (3) intervention/ practice regime; and (4) evaluation of outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders will be involved
2. Duration of the disease is more than 3 months.
3. Ischemic and hemorrhagic stroke will be included
4. Left sided hemiparesis
5. Hemiparetic patient, degree of spasticity for upper and lower limbs ranges from (grade 1+ : 2 ) according to modified Aschworth scale
6. Patient's age ranges from 45 to 60 years.
7. Patient's ability to stand independently for at least 5 minutes without the use of an assistive device.
8. Patients with sufficient cognitive abilities that enables them to understand and follow instructions (The Montreal Cognitive Assessment score >26) (Appendix II).
9. Body mass index for patients will not be more than 30.

Exclusion Criteria:

1. Neurological diseases that affect gait other than stroke (eg: Multiple sclerosis, Peripheral neuropathy, Parkinsonism etc.).
2. Musculoskeletal disorders such as severe arthritis, knee surgery, total hip joint replacement, lower limb fractures less than 6 months or contractures of fixed deformity, leg length discrepancy.
3. Cardiovascular problems (unstable angina, recent myocardial infarction within the last three months, congestive heart failure, significant heart valve dysfunction, or unstable hypertension) or pulmonary disorders.
4. Visual, auditory and speech problems.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic Gait Index | 1 year
  the DGI tests the ability of the participant to maintain walking balance while responding to different task demands, through various dynamic conditions. It is a useful test in individuals with vestibular and balance problems and those at risk of falls.
  It includes eight items, walking on level surfaces, changing speeds, head turns in horizontal and vertical directions, walking and turning 180 degrees to stop, stepping over and around obstacles, and stair ascent and descent.
  Each item is scored on a scale of 0 to 3, with 3 indicating normal performance and 0 representing severe impairment.
  The best possible score on the DGI is a 24
Berg Balance Scale | 1 year
  is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
Falls Efficacy Scale - International (FES-I) | 1 year
  It is a 16 item questionnaire, useful to the researchers and clinicians interested in fear of falling, with a score ranging from minimum 16 (no concern about falling) to maximum 64 (severe concern about falling)

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No